CLINICAL TRIAL: NCT05900947
Title: Presence of Environmental Pollutants in Human Carotid Atherosclerotic Plaques and Their Relationship With the Plaque Phenotype and Clinical Outcomes
Brief Title: Pollutants in the Atherosclerotic Plaque and Cardiovascular Events
Acronym: APAChE
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Cardarelli Hospital (Other); IRCCS Multimedica (Other)
Responsible Party: Principal Investigator, Raffaele Marfella, full professor, University of Campania Luigi Vanvitelli
Other Study IDs: 2704.2023
Record Dates: First submitted 2023-04-28; First posted 2023-06-13 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Carotid plaques
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: analysis of carotid atherosclerotic plaque — To assess the presence of air pollutants (benzene, toluene, xylene, and ethylbenzene) or of microplastics within tissues from atherosclerotic plaques by Chromatographic analyses.

SUMMARY:
Air pollution, microplastics and climate change pose serious public health risks. In recent years, air pollution has been associated with an increased risk of morbidity, all-cause mortality, cardio-respiratory-related mortality, and cancer.

A growing body of evidence has recently confirmed a direct association between particulate matter with an aerodynamic diameter less than or equal to 2.5 mm (PM2.5), Ozone (O3) and aromatic polycyclic hydrocarbons with all-cause mortality irrespective of social context and geographic or economic disparities, suggesting a causal relationship between the two factors.

The effects of air and environmental pollutants on public health have been observed also for short-term exposure to rapid increases in particulate matter.

High PM 2.5 values have also been associated with a higher rate of atherosclerosis and coronary artery disease expressed by high calcium score values, with the elderly, male and diabetic patients being at greater risk. To date, however, the pathophysiological basis of the relationship between air pollutants, and long-term events remains speculative, and there is no evidence that can correlate the concentration of environmental pollutants directly with anatomical-pathological and/or biomolecular alterations.

In this study the investigators will assess the presence and the burden of pollutants within the carotid plaques from patients undergoing carotid endarterectomy with pyrolysis-gas chromatography-mass spectrometry and electronic microscopy. Plaque stability will be explored trough molecular markers. Participants will be followed up for a composite of myocardial infarction, stroke, and all-cause mortality to evaluate whether the presence and the abundance of pollutants are associated with the development of the outcome through adjusted Cox regressions.

DETAILED DESCRIPTION:
Among patients with carotid stenosis (according to North American Symptomatic Carotid Endarterectomy Trial classification) enlisted to undergo carotid endarterectomy for extracranial high-grade (>70%) internal carotid artery stenosis, the investigators will enroll 300 consecutive patients with asymptomatic disease. All patients will undergo a baseline clinical examination, with computed tomography or MRI to assess cerebral lesions, and health records will be collected. Clinical variables will be measured with standard procedures after overnight fasting. Patients with evidence of heart failure, valvular defects, malignant neoplasms, or secondary causes of hypertension will be excluded.

Specimens of the portion of carotid bifurcation that showed maximum disease will be obtained from atherectomy and will be cut in two halves and frozen in liquid nitrogen or fixed in in 10% buffered formalin for subsequent analyses.

Plaque specimens will be then used to assess the presence and the amount of volatile organic compounds and microplastics through pyrolysis-gas chromatography-mass spectrometry.

To corroborate these findings, plaque specimens will be also observed with transmission electron microscopy to visually identify microplastics within the atheroma and obtain further evidence and structural insights.

Plaques will be also analysed through immunohistochemistry, ELISAs, and Western Blot to quantify inflammatory, i.e. NLRP3, caspase-1, IL-1β, IL-6, TNFα, NF-kB, and CD68, and plaque stability markers, i.e. MMP-9 and collagen, in order to explore whether the presence of microplastics is associated with a poorer plaque phenotype. The groups (composed post-hoc) of patients with polluted plaques vs non-polluted plaques will be compared for the expression of all these markers.

After carotid endarterectomy, patients will be followed-up and monitored for the incidence of a composite outcome constituted by non-fatal myocardial infarction, non-fatal stroke, and all-cause mortality, which represent the main and the only hard endpoint of the study.

Patients will be categorized (post-hoc) as having polluted plaques (having detectable levels of at least one pollutant) or non-polluted plaques. Cox regression analysis will be used to examine the association between the presence of microplastics and the incidence of the composite outcome, adjusted for age, sex, BMI, systolic and diastolic blood pressure, the prevalence of diabetes, dyslipidaemia, and smoking. Among those with polluted plaques, the abundance of pollutants, i.e. the sum, will be used to categorize patients into terciles. Cox models, adjusted for the same variables, will be run to explore the relationship between the burden of microplastics and the outcome. P values < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients with carotid stenosis (according to North American Symptomatic Carotid Endarterectomy Trial classification) enlisted to undergo carotid endarterectomy for extracranial high-grade (>70%) internal carotid artery stenosis.

Exclusion Criteria:

* All patients with clinical or laboratory evidence of heart failure, valvular defects, malignant neoplasms, or secondary causes of hypertension will be excluded from the study.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include the patients with carotid stenosis (according to North American Symptomatic Carotid Endarterectomy Trial classification) enlisted to undergo carotid endarterectomy for extracranial high-grade (>70%) internal carotid artery stenosis. The patients will be male and female subjects, with age > 18 and < 75 years. We will select patients with asymptomatic carotid disease. All patients will have a baseline clinical examination, and receive computed tomography or MRI to assess cerebral lesions, and previous health records will be evaluated. Clinical variables will be measured with standard procedures after overnight fasting. Patients with diabetes will be categorized according to the ADA criteria.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of a composite of myocardial infarction, stroke, and all-cause mortality in patients with polluted vs non-polluted plaques | 24 months
  Patients will be categorized (post-hoc) as having polluted plaques (having detectable levels of at least one microplastics) or non-polluted plaques. Cox regression analysis will be used to examine the association between the presence of pollutants (yes/no) and the incidence of the composite outcome, adjusted for age, sex, BMI, systolic and diastolic blood pressure, the prevalence of diabetes, dyslipidaemia, and smoking.

SECONDARY OUTCOMES:
Incidence of a composite of myocardial infarction, stroke, and all-cause mortality according to terciles of pollutants burden | 24 months
  Among those with polluted plaques, the abundance of pollutants, i.e. the sum, will be used to categorize patients into terciles. Cox models, adjusted for the same variables, will be run to explore the relationship between the burden of microplastics and the outcome. P values < 0.05 will be considered statistically significant.

OTHER OUTCOMES:
Comparison of plaque stability markers between polluted and non-polluted plaques | 12 months
  Plaques will be also analysed through immunohistochemistry to quantify plaque stability markers (in arbitrary units), i.e. MMP-9 and collagen, in order to explore whether the presence of pollutants is associated with a poorer plaque phenotype. The groups (composed post-hoc) of patients with polluted plaques vs non-polluted plaques will be compared for the expression of all these markers through t test or Mann-Whitney U test, according to the distribution of the variables.
Comparison of inflammatory markers between polluted and non-polluted plaques | 12 months
  Plaques will be also analysed through Western Blot to quantify inflammatory markers (in arbitrary units), i.e. NLRP3, caspase-1, IL-1β, IL-6, TNFα, NF-kB, and CD68, in order to explore whether the presence of pollutants is associated with a poorer plaque phenotype. The groups (composed post-hoc) of patients with polluted plaques vs non-polluted plaques will be compared for the expression of all these markers through t test or Mann-Whitney U test, according to the distribution of the variables.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Marfella, MD,PhD, Principal Investigator — Università della Campania Vanvitelli; Celestino Sardu, MD, Study Chair — Università degli Studi della Campania; Francesco Prattichizzo, PhD, Study Chair — IRCCS Multimedica
Locations (1):
- Celestino Sardu, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perera F, Nadeau K. Climate Change, Fossil-Fuel Pollution, and Children's Health. N Engl J Med. 2022 Jun 16;386(24):2303-2314. doi: 10.1056/NEJMra2117706. No abstract available. PMID 35704482
- [Background] Lim SS, Vos T, Flaxman AD, Danaei G, Shibuya K, Adair-Rohani H, Amann M, Anderson HR, Andrews KG, Aryee M, Atkinson C, Bacchus LJ, Bahalim AN, Balakrishnan K, Balmes J, Barker-Collo S, Baxter A, Bell ML, Blore JD, Blyth F, Bonner C, Borges G, Bourne R, Boussinesq M, Brauer M, Brooks P, Bruce NG, Brunekreef B, Bryan-Hancock C, Bucello C, Buchbinder R, Bull F, Burnett RT, Byers TE, Calabria B, Carapetis J, Carnahan E, Chafe Z, Charlson F, Chen H, Chen JS, Cheng AT, Child JC, Cohen A, Colson KE, Cowie BC, Darby S, Darling S, Davis A, Degenhardt L, Dentener F, Des Jarlais DC, Devries K, Dherani M, Ding EL, Dorsey ER, Driscoll T, Edmond K, Ali SE, Engell RE, Erwin PJ, Fahimi S, Falder G, Farzadfar F, Ferrari A, Finucane MM, Flaxman S, Fowkes FG, Freedman G, Freeman MK, Gakidou E, Ghosh S, Giovannucci E, Gmel G, Graham K, Grainger R, Grant B, Gunnell D, Gutierrez HR, Hall W, Hoek HW, Hogan A, Hosgood HD 3rd, Hoy D, Hu H, Hubbell BJ, Hutchings SJ, Ibeanusi SE, Jacklyn GL, Jasrasaria R, Jonas JB, Kan H, Kanis JA, Kassebaum N, Kawakami N, Khang YH, Khatibzadeh S, Khoo JP, Kok C, Laden F, Lalloo R, Lan Q, Lathlean T, Leasher JL, Leigh J, Li Y, Lin JK, Lipshultz SE, London S, Lozano R, Lu Y, Mak J, Malekzadeh R, Mallinger L, Marcenes W, March L, Marks R, Martin R, McGale P, McGrath J, Mehta S, Mensah GA, Merriman TR, Micha R, Michaud C, Mishra V, Mohd Hanafiah K, Mokdad AA, Morawska L, Mozaffarian D, Murphy T, Naghavi M, Neal B, Nelson PK, Nolla JM, Norman R, Olives C, Omer SB, Orchard J, Osborne R, Ostro B, Page A, Pandey KD, Parry CD, Passmore E, Patra J, Pearce N, Pelizzari PM, Petzold M, Phillips MR, Pope D, Pope CA 3rd, Powles J, Rao M, Razavi H, Rehfuess EA, Rehm JT, Ritz B, Rivara FP, Roberts T, Robinson C, Rodriguez-Portales JA, Romieu I, Room R, Rosenfeld LC, Roy A, Rushton L, Salomon JA, Sampson U, Sanchez-Riera L, Sanman E, Sapkota A, Seedat S, Shi P, Shield K, Shivakoti R, Singh GM, Sleet DA, Smith E, Smith KR, Stapelberg NJ, Steenland K, Stockl H, Stovner LJ, Straif K, Straney L, Thurston GD, Tran JH, Van Dingenen R, van Donkelaar A, Veerman JL, Vijayakumar L, Weintraub R, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams W, Wilson N, Woolf AD, Yip P, Zielinski JM, Lopez AD, Murray CJ, Ezzati M, AlMazroa MA, Memish ZA. A comparative risk assessment of burden of disease and injury attributable to 67 risk factors and risk factor clusters in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2224-60. doi: 10.1016/S0140-6736(12)61766-8. PMID 23245609
- [Background] Di Q, Wang Y, Zanobetti A, Wang Y, Koutrakis P, Choirat C, Dominici F, Schwartz JD. Air Pollution and Mortality in the Medicare Population. N Engl J Med. 2017 Jun 29;376(26):2513-2522. doi: 10.1056/NEJMoa1702747. PMID 28657878
- [Background] Bevan GH, Al-Kindi SG, Brook RD, Munzel T, Rajagopalan S. Ambient Air Pollution and Atherosclerosis: Insights Into Dose, Time, and Mechanisms. Arterioscler Thromb Vasc Biol. 2021 Feb;41(2):628-637. doi: 10.1161/ATVBAHA.120.315219. Epub 2020 Dec 17. PMID 33327745
- [Derived] Marfella R, Prattichizzo F, Sardu C, Fulgenzi G, Graciotti L, Spadoni T, D'Onofrio N, Scisciola L, La Grotta R, Frige C, Pellegrini V, Municino M, Siniscalchi M, Spinetti F, Vigliotti G, Vecchione C, Carrizzo A, Accarino G, Squillante A, Spaziano G, Mirra D, Esposito R, Altieri S, Falco G, Fenti A, Galoppo S, Canzano S, Sasso FC, Matacchione G, Olivieri F, Ferraraccio F, Panarese I, Paolisso P, Barbato E, Lubritto C, Balestrieri ML, Mauro C, Caballero AE, Rajagopalan S, Ceriello A, D'Agostino B, Iovino P, Paolisso G. Microplastics and Nanoplastics in Atheromas and Cardiovascular Events. N Engl J Med. 2024 Mar 7;390(10):900-910. doi: 10.1056/NEJMoa2309822. PMID 38446676